CLINICAL TRIAL: NCT05003726
Title: Comparative Effectiveness of Non-pharmacological Treatment and Pharmacological Treatment for Non-acute Lumbar Disc Herniation : a Multi-centered, Pragmatic Randomized Controlled, Parallel-grouped Pilot Study
Brief Title: Non-pharmacological Treatment and Pharmacological Treatment for Non-acute Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Principal Investigator, Kyoung Sun Park, Chief, clinical study center, Jaseng Hospital of Korean Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2021-07
Record Dates: First submitted 2021-08-11; First posted 2021-08-12 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Lumbar Disc Herniation; Radiculopathy Lumbar
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-pharmacological group including KM (Experimental): Non-pharmacological treatment including Korean medicine will be implemented to the participants for total 8 weeks. This is a pragmatic clinical trial, and the specific intervention will be determined according to the physician's choice. intervention data will be recorded in the case report form.
  Interventions: Procedure: non-pharmacological treatment
- Pharmacological group (Active Comparator): Pharmacological treatment will be implemented to the participants for total 8 weeks. This is a pragmatic clinical trial, and the specific intervention will be determined according to the physician's choice. intervention data will be recorded in the case report form.
  Interventions: Procedure: pharmacological treatment

INTERVENTIONS:
Procedure: non-pharmacological treatment — This is a pragmatic setting, and specific intervention is not determined prior to the study. Non-pharmacological treatment including Korean medicine, such as acupuncture, electroacupuncture and chuna, etc, will be chosen by professional physician according to the medical condition of each subject.
  Arms: Non-pharmacological group including KM
Procedure: pharmacological treatment — This is a pragmatic setting, and specific intervention is not determined prior to the study. The pharmacological treatment will be chosen by professional physician according to the medical condition of each subject.
  Arms: Pharmacological group

SUMMARY:
This study is a 2-armed parallel, multi-centered, pragmatic clinical trial that compares the comparative effectiveness of non-pharmacological treatment and pharmacological treatment for non-acute lumbar disc herniation.

DETAILED DESCRIPTION:
This study is a multi-centered, pragmatic clinical trial that compares the comparative effectiveness of non-pharmacological treatment and pharmacological treatment for non-acute lumbar disc herniation. The participants who voluntarily signed informed consent will be randomly assigned in 1:2 ratio to non-pharmacological group and pharmacological group and will receive the 8 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Numeric rating scale (NRS) score of radiating pain or low back pain 5 or more for recent 3 serial days.
2. Onset time of radiating pain occurred 3 months before enrollment.
3. Radiologically diagnosed with lumbar disc herniation in lumbar spine magnetic resonance imaging (L-spine MRI), which can explain lower extremity radiation pain and back pain
4. 19-69 years old
5. participants who agreed and signed informed consent form

Exclusion Criteria:

1. Spine metastasis of cancer, acute fracture of spine, or spine dislocation
2. Progressive neurologic deficits or severe neurologic deficits
3. Soft tissue diseases that can induce low back pain(ie. cancer, fibromyalgia, rheumatoid arthritis, gout,etc)
4. Presence of chronic underlying disease which can interfere the efficacy or interpretation (ie. stroke, myocardial infarct, kidney disease, dementia, diabetic neuropathy, epilepsy, etc)
5. Concurrent use of steroids, immunosuppressants, orpsychotropic medications or any other medication that can interrupt the study result
6. Hemorrhagic disease, severe diabetes or taking anticoagulant drug
7. Participants who took NSAIDs within 1 week
8. Pregnant or lactating women
9. Participants who had undergone lumbar surgery within 3 months
10. Participants who had participated in other clinical trial within 1 month, or have plan for participation in other trial during follow up period of this trial
11. Participants who can not write informed consent
12. Participants who is difficult to participate in the trial according to investigator's decision

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index (ODI) | week 1, 5, 9, 14, 27
  ODI is a functional disability questionnaire. The possible range of eachitem score is 0 to 5. Total score range is 0 (better outcome) to 100 (worse outcome)

SECONDARY OUTCOMES:
Numeric rating scale (NRS) of low back pain | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 14, 27
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Visual analogue scale (VAS) of low back pain and radiating pain in lower extermities | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 14, 27
  Visual analogue scale of low back pain and radiating leg pain, minimum 0 to maximum 100,which is a higher score means a worse outcome.
Numeric rating scale (NRS) of radiating pain in lower extremities | week -1, 1, 2, 3, 4, 5, 6, 7, 8, 9, 14, 27
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Patient global impression of change (PGIC) | week 9, 14, 27
  Participants rate the global impression of improvement after treatment on a 7-point Likert scale.
Short form-12 health survey version 2 (SF-12 v2) | week 1, 5, 9, 14, 27
  The SF-12 consists of 12 questions across 8 domains, and higher scores indicate better health-related quality of life.
EuroQol-5 Dimension (EQ-5D-5L) | week 1, 5, 9, 14, 27
  The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about)
Credibility and Expectancy | week -1
  To evaluate participants' expectations for treatment, the nine-point scale(Likert scale) is used to evaluate them. During the screening visit, the candidates will choose their scores in response to the question, "How much do you think non-drug therapy, including Korean medical treatment, or medication will relieve your symptoms?" (1 = not at all, 5 = somewhat, and 9 = very much)
Evaluation question | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 14, 27
  Use a questionnaire that measures official unofficial medical expenses, non-medical expenses, time costs, and productivity loss costs developed separately to measure cost items. Informal medical expenses, such as purchasing pars or medical devices, include transportation, patient time, transportation, patient time, and nursing costs are non-medical expenses. Productivity loss costs refer to the cost of economic loss caused by the disease itself or by the inability to participate in labor due to premature death from the disease. To calculate the cost of productivity loss, we will use the Work Productivity and Activity Impairment questionnair (WPAI) to convert it into cost-effectiveness analysis.
Drug Consumption | week -1, 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 14, 27
  The type and dose of prescribed drugs or relief drugs due to the active history of drugs taken during the study period are observed through a questionnaire when visiting the study subjects. Other than the medication you are taking, physical therapy, injection therapy, etc. should be recorded in the number of times.
Adverse events | week -1, 1, 2, 3, 4, 5, 6, 7, 8, 9, 14, 27
  Safety will be verified by comparing the occurrence of adverse events between the two groups. The researcher evaluates each treatment method and its adverse events on a six-step scale according to the WHO-UMC UMC causality assessment system (1=definitive linked, 2=provocatively linked, 4=probably not related, 5=definitive not related, 5=definitive not related to the study), and all adverse events are classified into three stages by the Spilker taxonomy (Mild(1)): If treatment is not required and does not significantly impair the normal life function, Moderate(2): may significantly impair normal life function, and may require treatment, and Severe(3): severe adverse events require high treatment, and side effects remain.

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Sun Park, Ph.D, Principal Investigator — Jaseng Hospital of Korean Medicine
Locations (4):
- South Korea (4):
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon
  - Jaseng Hospital of Korean Medicine, Seoul

IPD SHARING:
Plan to Share IPD: No